CLINICAL TRIAL: NCT00002548
Title: Standard Dose Versus Myeloablative Therapy for Previously Untreated Symptomatic Multiple Myeloma, A Phase III Intergroup Study
Brief Title: SWOG-9321 Melphalan, TBI, and Transplant vs Combo Chemo in Untreated Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWOG-9321; SWOG-9321 (Other: SWOG); CLB-9312 (Other: CALGB); E-S9321 (Other: ECOG); INT-0141 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-08-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Interferon-alpha; Carmustine; Cyclophosphamide; Dexamethasone; Steroids; Calcium Dobesilate; Doxorubicin; Melphalan; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HDCTX and PBSC (Active Comparator): High dose chemotherapy with peripheral blood stem cells
  High dose chemotherapy with peripheral blood stem cells IND (q 5 weeks): vincristine 0.5 mg/d cont IV D1-4; adriamycin 10mg/m2/d cont IV D1-4; dex 40 mg/d PO or IVPB D1-4, 9-12, 17-20
  2nd Reg: cyclophosphamide 1.5g/m2 IV over 1 hr every 3 hrs x 3 (4.5g/m2 total); MESNA 4.5 g/m2 24 hr IV start with cyclo; GCSF 0.25 mg/m2/d SQ; PBSC collection
  Chemo: vincristine 1.2 mg/m2 IV D1, BCNU 20 mg/m2 IV D1, melphalan 8 mg/m2 PO D1-4, cyclophosphamide 400 mg/m2 IV D1, prednisone 40 mg/m2 PO D1-7
  Interventions: Drug: doxorubicin hydrochloride; Drug: melphalan; Drug: prednisone; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation
- HDCTX with PBSC and Autologous BMT (Experimental): High dose chemotherapy with peripheral blood stem cells and autologous bone marrow transplant
  High dose chemotherapy with peripheral blood stem cells and autologous bone marrow transplant
  High dose chemotherapy with peripheral blood stem cells IND (q 5 weeks): vincristine 0.5 mg/d cont IV D1-4; adriamycin 10mg/m2/d cont IV D1-4; dex 40 mg/d PO or IVPB D1-4, 9-12, 17-20
  2nd Reg: cyclophosphamide 1.5g/m2 IV over 1 hr every 3 hrs x 3 (4.5g/m2 total); MESNA 4.5 g/m2 24 hr IV start with cyclo; GCSF 0.25 mg/m2/d SQ; PBSC collection
  Auto Trans: Mel 140mg/m2 IV D-5; TBI 150cGy D-4, -3, -2, -1; infusion D0
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: melphalan; Drug: prednisone; Procedure: allogeneic bone marrow transplantation; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- HDCTX with PBSC and interferon (Experimental): High dose chemotherapy with peripheral blood stem cells and interferon
  Experimental: HDCTX with PBSC and interferon High dose chemotherapy with peripheral blood stem cells and interferon
  High dose chemotherapy with peripheral blood stem cells IND (q 5 weeks): vincristine 0.5 mg/d cont IV D1-4; adriamycin 10mg/m2/d cont IV D1-4; dex 40 mg/d PO or IVPB D1-4, 9-12, 17-20
  2nd Reg: cyclophosphamide 1.5g/m2 IV over 1 hr every 3 hrs x 3 (4.5g/m2 total); MESNA 4.5 g/m2 24 hr IV start with cyclo; GCSF 0.25 mg/m2/d SQ; PBSC collection
  Chemo: vincristine 1.2 mg/m2 IV D1, BCNU 20 mg/m2 IV D1, melphalan 8 mg/m2 PO D1-4, cyclophosphamide 400 mg/m2 IV D1, prednisone 40 mg/m2 PO D1-7
  IFN: IFN 3 million units/m2 MWF SQ
  Interventions: Biological: recombinant interferon alfa; Drug: doxorubicin hydrochloride; Drug: melphalan; Drug: prednisone; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation
- HDCTX with PBSC and transplant plus IFN (Experimental): High dose chemotherapy with peripheral blood stem cells and autologous bone marrow transplant plus alpha interferon
  Experimental: HDCTX with PBSC and transplant plus IFN High dose chemotherapy with peripheral blood stem cells and autologous bone marrow transplant plus alpha interferon
  High dose chemotherapy with peripheral blood stem cells IND (q 5 weeks): vincristine 0.5 mg/d cont IV D1-4; adriamycin 10mg/m2/d cont IV D1-4; dex 40 mg/d PO or IVPB D1-4, 9-12, 17-20
  2nd Reg: cyclophosphamide 1.5g/m2 IV over 1 hr every 3 hrs x 3 (4.5g/m2 total); MESNA 4.5 g/m2 24 hr IV start with cyclo; GCSF 0.25 mg/m2/d SQ; PBSC collection
  Trans: Mel 140mg/m2 IV D-5; TBI 150cGy D-4, -3, -2, -1; infusion D0
  IFN: 3 million units/m2 MWF SQ
  Interventions: Biological: recombinant interferon alfa; Drug: carmustine; Drug: cyclophosphamide; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: melphalan; Drug: prednisone; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: recombinant interferon alfa — 3 million units/m2 SQ Monday-Wednesday
  -Friday (3 times a week)
  Other Names: IFN, alpha interferon
  Arms: HDCTX with PBSC and interferon; HDCTX with PBSC and transplant plus IFN
Drug: carmustine — 20 mg/m2 I.V. day 1 q 35 days
  Other Names: BCNU
  Arms: HDCTX with PBSC and Autologous BMT; HDCTX with PBSC and transplant plus IFN
Drug: cyclophosphamide — 1.5 g/m2 in 100 ml of D5W, IV intravenously over 1 hour every 3 hour x 3 (total dose 4.5 g/m2)
  Other Names: cytoxan
  Arms: HDCTX with PBSC and Autologous BMT; HDCTX with PBSC and transplant plus IFN
Drug: dexamethasone — 40 mg/day PO or IVPB days 1-4, 9-12, 17-20 q 5 weeks
  Other Names: steroid, decadron
  Arms: HDCTX with PBSC and Autologous BMT; HDCTX with PBSC and transplant plus IFN
Drug: doxorubicin hydrochloride — 10 mg/m2/day continuous 1 - 4 q 5 weeks
  Other Names: Adriamycin
Drug: melphalan — 140 mg/m2 is given IV within 30 minutes of constitution on Day -5
Drug: prednisone — 40 mg/m2 PO days 1-7 q 35 days
Drug: vincristine sulfate — 0.5 mg/day continuous 1 - 4 q 5 weeks
  Arms: HDCTX and PBSC; HDCTX with PBSC and interferon
Procedure: allogeneic bone marrow transplantation — day 0
  Arms: HDCTX with PBSC and Autologous BMT
Procedure: autologous bone marrow transplantation — day 0
  Arms: HDCTX with PBSC and Autologous BMT; HDCTX with PBSC and transplant plus IFN
Procedure: peripheral blood stem cell transplantation — day 0
Radiation: radiation therapy — administered in fractionated doses of 150 cGy, 6 - 10 hours apart bid, on Days -4, -3, -2, and -1 (Total 1,200 cGy)
  Arms: HDCTX with PBSC and Autologous BMT; HDCTX with PBSC and transplant plus IFN

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy and radiation therapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and radiation therapy and kill more cancer cells. It is not yet known which treatment regimen is more effective for multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of melphalan, total-body irradiation, and peripheral stem cell transplantation with that of combination chemotherapy in treating patients who have previously untreated multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare tumor cytoreduction achieved with VBMCP (vincristine/carmustine/melphalan/cyclophosphamide/prednisone) vs myeloablative melphalan (L-PAM) and total-body irradiation (TBI) with peripheral blood stem cell (PBSC) rescue in symptomatic myeloma patients with stable or responding disease after induction therapy with VAD (vincristine/doxorubicin/dexamethasone) followed by high dose cyclophosphamide plus filgrastim (G-CSF).
* Compare the efficacy of interferon alfa vs no maintenance therapy in those patients achieving at least 75% cytoreduction to either VBMCP or myeloablative therapy with PBSC rescue.
* Assess allogeneic bone marrow transplantation following the same myeloablative regimen of L-PAM/TBI in patients up to age 55 with an HLA-compatible, MLC-nonreactive donor. (As of 8/1/97, permanent partial closure)
* Determine whether myeloablative therapy with PBSC rescue can extend the duration of survival by 33% compared to results from standard dose VBMCP.
* Evaluate the toxic effects and possible long term side effects, including development of myelodysplastic disease and/or acute myeloblastic leukemia, associated with these treatments.

OUTLINE: This is a randomized study. Patients are registered at 5 different points, with stratification occurring at some of these registrations.

* Registration I: Induction I
* Registration II: Induction II. Patients are stratified according to stage of disease (I/II vs IIIA vs IIIB), beta-2 microglobulin at diagnosis (less than 6 micrograms/mL vs at least 6 micrograms/mL), and response to Induction I (75-100% regression vs 50-74% regression vs less than 50% regression vs not applicable).
* Registration III: Patients are randomized to allogeneic bone marrow transplant (BMT) (this arm closed as of 8/1/97) or autologous BMT. Patients are stratified according to treatment received (high dose cyclophosphamide (CTX) and peripheral blood stem cells (PBSC) prior to autologous BMT vs prior to chemotherapy) and beta-2 microglobulin at this registration (less than 2 micrograms/mL vs no greater than 3 micrograms/mL vs unknown).
* Registration IV: Patients are randomized to maintenance therapy or no further therapy. Those patients who are randomized to maintenance therapy are stratified according to treatment (autologous BMT vs chemotherapy vs chemotherapy followed by autologous BMT) and response to treatment (75-99% regression vs complete response).
* Registration V: Patients receive autologous BMT as in registration III. Patients are stratified according to prior best response (50% or better vs less than 50% vs not applicable), duration of chemotherapy (at least 6 months vs less than 6 months), and progression after therapy (chemotherapy vs interferon alfa vs observation).
* Induction I: Patients receive vincristine IV and doxorubicin IV by continuous infusion on days 1-4 and dexamethasone IV or orally on days 1-4, 9-12, and 17-20. Treatment repeats every 5 weeks for up to 4 courses. Patients with progressive disease after 2 courses proceed to PBSC stimulation/harvest.

Allogeneic BMT arm is permanently closed as of 8/1/97.

* Autologous BMT: Therapy begins 4-8 weeks following high dose cyclophosphamide. Patients receive melphalan IV over 1 hour on day -5 and total body irradiation twice a day on days -4 to -1. PBSC are reinfused on day 0. G-CSF SQ is administered beginning on day 1 until blood counts recover.
* Chemotherapy: Patients receive vincristine IV, carmustine IV, and cyclophosphamide IV on day 1, oral melphalan on days 1-4, and oral prednisone on days 1-7. Treatment repeats every 5 weeks for at least 12 months.

Patients who have at least a 75% response to autologous BMT or chemotherapy are randomized to maintenance vs no further therapy. Patients who progress on chemotherapy proceed to autologous BMT (registration V).

* Maintenance therapy: Therapy begins between 5 and 12 weeks after PBSC rescue. Patients receive interferon alfa SQ three times a week. Treatment continues for 4 years in the absence of disease progression or unacceptable toxicity.

Patients who progress on chemotherapy undergo an autologous BMT within 8 weeks after the last course of chemotherapy.

Patients who are randomized to receive no further therapy are observed for 1 year.

PROJECTED ACCRUAL: A total of 500 patients will be randomized over about 4 years to autologous transplantation vs chemotherapy as follows: about 250 patients/year will be accrued for induction of whom 200 will achieve at least stable disease, 125 will be randomized, and 15 will have a suitable donor for allogeneic transplant (as of 8/1/97, allogeneic arm of study is closed). Approximately 300 patients are expected to be randomized to maintenance vs no further therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed, active multiple myeloma of any stage requiring treatment

  * Smoldering myeloma (Durie-Salmon stage I) must have a 25% or greater increase in M component levels and/or Bence-Jones protein excretion or development of symptoms
* Quantifiable M component of IgG, IgA, IgD, IgE, and/or urinary kappa or lambda light chain (Bence-Jones protein) excretion required

  * Plasmacytosis of at least 30% allowed for non-secretory disease or secretory disease without quantifiable protein
  * IgM peaks excluded
* Evaluation of siblings as potential allogeneic bone marrow transplant donors required for patients 55 years of age and younger (As of 8/1/97, permanently closed)

  * HLA followed by DR and MLC testing required
* Renal failure, even on dialysis, eligible provided:

  * Cause is attributed to myeloma (Bence-Jones protein or hypercalcemia)
  * Duration does not exceed 2 months
* If medically appropriate, the following conditions should be treated prior to registration:

  * Pathologic fractures
  * Pneumonia at diagnosis
  * Hyperviscosity with shortness of breath

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Performance status:

* SWOG 0-2 (SWOG 3 or 4 based solely on bone pain allowed)

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* See Disease Characteristics

Cardiovascular:

* Normal ejection fraction by ECHO or MUGA
* No myocardial infarction within 6 months
* No unstable angina
* No difficult to control congestive heart failure
* No uncontrolled hypertension
* No difficult to control arrhythmias
* No history of chronic cerebral vascular accident

Pulmonary:

* No history of chronic obstructive or restrictive pulmonary disease
* Pulmonary function studies and DLCO at least 50% of predicted except for demonstrated myeloma involvement on bronchoscopy and/or open lung biopsy

Other:

* No uncontrolled diabetes
* No significant comorbid medical condition
* No uncontrolled, life-threatening infection
* No prior malignancy within 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No prior malignancy treated with cytotoxic drugs used on this protocol
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy except local radiotherapy provided the following cumulative dose limits for prior dose plus potential TBI dose on protocol are not exceeded:

  * Less than 5,000 cGy to bone
  * Less than 4,000 cGy to mediastinum, heart, small bowel, brain, and spinal cord
  * Less than 2,000 cGy to the liver
  * Less than 1,500 cGy to the kidney and lungs

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 1994-01; Primary Completion 2003-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
survival | 3 years from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, Study Chair — University of Arkansas; Kenneth C. Anderson, MD, Study Chair — Dana-Farber Cancer Institute; Robert A. Kyle, MD, Study Chair — Mayo Clinic
Locations (34):
- United States (34):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin

REFERENCES:
- [Background] van Ness BG, Ramos C, Kumar V, et al.: Analytical approaches for the BOAC SNP panel association with progression free survival in myeloma. [Abstract] Blood 112 (11): A-2715, 2008.
- [Background] Crowley JJ, McCoy J, LeBlanc M, et al.: Extreme regression: a statistical technique for finding good or poor prognostic groups, illustrated using myeloma patient data from Intergroup trial S9321. [Abstract] Blood 104 (11): A-5202, 2004.
- [Background] Greipp PR, Kumar S, Blood EA, et al.: A simple classification to identify poor-risk untreated myeloma. [Abstract] Blood 100 (11 Pt 1): A-2351, 598a, 2002.
- [Background] Tian E, Bumm K, Xiao Y, et al.: A protocol for triple color interphase FISH on archived bone marrow biopsies from myeloma prepared with precipitating fixatives. [Abstract] Blood 96 (11 pt 1): A-665, 155a, 2000.
- [Background] Rajkumar V, Leong T, Fonseca R, et al.: Bone marrow angiogenesis has prognostic value in multiple myeloma: an Eastern Cooperative Oncology Group study. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A68, 19a, 1999.
- [Background] Rimsza LM, Campbell K, Dalton WS, Salmon S, Willcox G, Grogan TM. The major vault protein (MVP), a new multidrug resistance associated protein, is frequently expressed in multiple myeloma. Leuk Lymphoma. 1999 Jul;34(3-4):315-24. doi: 10.3109/10428199909050956. PMID 10439368
- [Result] Barlogie B, Kyle RA, Anderson KC, Greipp PR, Lazarus HM, Hurd DD, McCoy J, Moore DF Jr, Dakhil SR, Lanier KS, Chapman RA, Cromer JN, Salmon SE, Durie B, Crowley JC. Standard chemotherapy compared with high-dose chemoradiotherapy for multiple myeloma: final results of phase III US Intergroup Trial S9321. J Clin Oncol. 2006 Feb 20;24(6):929-36. doi: 10.1200/JCO.2005.04.5807. Epub 2006 Jan 23. PMID 16432076
- [Result] Van Ness BG, Crowley JC, Ramos C, et al.: SNP genotypes show association with common toxicities during both VAD induction and high dose melphalan with autologous transplant support in intergroup trial S9321 for myeloma: from the Bank on a Cure. [Abstract] Blood 106 (11): A-3488, 2005.
- [Result] Crowley J, Fonseca R, Greipp P, et al.: Comparable survival in newly diagnosed multiple myeloma (MM) after VAD induction with high dose therapy using melphalan 140mg/m2 + TBI 12 Gy (MEL+TBI) versus standard therapy with VBMCP and no benefit from interferon (IFN) maintenance: final clinical results of intergroup trial S9321 in the context of IFM 90 and MRC VII trials. [Abstract] Blood 104 (11): A-539, 2004.
- [Result] Santana-Davila R, Crowley J, Durie B, et al.: Genetic polymorphisms associated with clinical outcome in the intergroup trial S9321, comparing high dose therapy with standard dose therapy for myelomaon, on behalf of ECOG, SWOG, CALGB, and the Bank on a Cure. [Abstract] Blood 104 (11): A-1495, 2004.
- [Result] Lee CK, McCoy J, Anderson KC, et al.: Long-term follow-up of previously untreated symptomatic myeloma patients treated with myeloablative therapy and sibling-matched allogeneic transplantation of the SWOG study 9321. [Abstract] Blood 100 (11 pt 1): A-1644, 2002.
- [Result] Greipp PR, Jacobson JL, Crowley JJ, et al.: BETA 2 microglobulin (beta 2M) and plasma cell labeling index (PCLI) constitute a strong prognostic index in the SWOG intergroup transplant trial S9321: observations on gender and age. [Abstract] Blood 96 (11 pt 1): A-653, 152a, 2000.
- [Result] Desika R, Salmon S, Anderson K, et al.: Planned melphalan-total body irradiation (MEL-TBI) - based allogeneic transplantation for multiple myeloma (MM) up to age 55: an intergroup experience (CALGB, ECOG and SWOG) under the auspices of the Southwest Oncology Group (SWOG 9321). [Abstract] Blood 94 (10 Pt 1): A-1546, 346a, 1999.
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675